CLINICAL TRIAL: NCT06406283
Title: Active Young, Healthy Mind: Strategies for Brain Health and Psychological Well-being in Young Adults: A Randomized Mixed-method Study With and Without Virtual Reality (VR) (YoungFitT: Young Fitness Technology)
Brief Title: Active Young, Healthy Mind. The YoungFitT Project
Acronym: YoungFitT
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Barcelona (Other)
Collaborators: University Ramon Llull (Other); ICREA Academia (Unknown); Institut de Neurociències de la Universitat de Barcelona (Unknown); Institut de Recerca Sant Joan de Déu (CERCA center) (Unknown); EventLab (Unknown); INEFC (Unknown); Nirakara Lab (Industry); Adventhealth Research Institute, Neuroscience (Unknown); University of Murdock (Unknown)
Responsible Party: Principal Investigator, Maria Mataro Serrat, Principal Investigator, University of Barcelona
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: UB; PID2022-137776OB-100 (Other Grant/Funding Number: Ministerio de Ciencia e Innovación (Gobierno de España)])
Record Dates: First submitted 2024-04-10; First posted 2024-05-09 (Actual); Last update posted 2024-05-09 (Actual); Status verified 2024-05

CONDITIONS: University Students
Keywords: Well-being; Physical exercise; Qigong; Mindfulness; Neuroimaging; Intervention; Randomization; Cognition; Virtual environment
MeSH Terms: conditions — Motor Activity | interventions — Qigong

STUDY DESIGN:
Intervention Model Description: In Study 1: 174 participants, all of them university students aged 18 to 25 years old, are randomly assigned to one of three arms: The first group (n=58) receives HIFT. The second group (n=58) receives Qigong. Finally, the third group (n=58) receives MBSR.
  In Study 1: 45 participants, all of them university students aged 18 to 25 years old, are randomly assigned to one of three arms: The first group (n=15) receives HIFT-VR. The second group (n=15) receives Qigong-VR. Finally, the third group (n=15) receives MBSR-VR.
Who Masked: Investigator, Outcomes Assessor
Masking Description: The randomization sequence is concealed (blinded) from research personnel, so that the investigators are not aware of whether a particular subject has been randomized to one of the intervention groups or to the active control group.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- High-Intensity Functional Training (HIFT) Group (Experimental)
  Interventions: Behavioral: High-Intensity Functional Training (HIFT)
- Mindfulness Group (Experimental)
  Interventions: Behavioral: Mindfulness-Based Stress Reduction Program (MBSR)
- Qigong Group (Experimental)
  Interventions: Behavioral: Qigong

INTERVENTIONS:
Behavioral: High-Intensity Functional Training (HIFT) — This intervention will include three sessions per week: two group 60-minute zoom online synchronous sessions guided by experts and one individual autonomous session (a repetition of a chosen session of that week).
  The training protocol will be designed based on Cross-Training workouts, emphasizing high-intensity interval training combined with functional resistance-training movements.
  Arms: High-Intensity Functional Training (HIFT) Group
Behavioral: Mindfulness-Based Stress Reduction Program (MBSR) — This intervention follows the official MBSR program designed by Jon Kabat-Zinn with some adaptations, as we did in Bermudo-Gallaguet, et al. (2022). The intervention will occur three days a week, including one 120-minute online synchronous session and two 20-40 min individual practices. The intensity of physical exercise will be adjusted to personal baseline characteristics.
  Arms: Mindfulness Group
Behavioral: Qigong — This intervention will include three sessions per week: two group 60-minute zoom online synchronous sessions guided by experts and one individual autonomous session (a repetition of a chosen session of that week).
  The program includes the Baduanjin sequence, considered one of the most ancient and beneficial forms for physical and mental health within the Qigong tradition.
  Arms: Qigong Group

SUMMARY:
The main objective of YoungFitT Project is to study the effect and neuro-psycho-biological mechanisms of mind and body interventions, also in the form of virtual reality (VR), on brain health, cognitive and psychological well-being of college students. The investigators have adopted an inter and multidisciplinary and multimodal approach to provide a more integrative perspective using cognitive, psychological, biochemical, and neuroimaging measurements. The investigators hypothesize that all three interventions Mindfulness-Based Stress Reduction (MBSR), Qigong, and High-Intensity Functional Training (HIFT) will produce gains in cognitive functions and psychological well-being at three months compared to baseline. Also, all three interventions will induce changes in the microbiota and brain structure and function. Finally, using a VR environment for these interventions will provide greater adherence and cognitive and psychological well-being benefits than conventional training.

DETAILED DESCRIPTION:
The YoungFitT Project is a multicentric, prospective, parallel, single-blinded, three-arm, mixed-method randomized clinical trial with a sample of 219 participants. All of participants are university students aged 18 to 25 years old and will be randomized through a computer-generated allocation sequence with a 1:1:1 ratio and stratified by sex.

The YoungFitT Project is divided into two Studies:

Study 1: Online-based mind and body interventions. A total of 174 eligible university students will be randomized into three groups of HIFT, Qigong and MBSR (n=58). All interventions last 12 weeks.

Study 2: VR-based mind and body interventions. A total of 45 eligible university students will be randomized into three groups of HIFT-VR, Qigong-VR and MBSR-VR (n=15). All interventions last 12 weeks.

In both, within two weeks before and after the interventions, medical, cognitive, and physical assessments will be performed. Neuroimaging and biological samples will be collected in Study 1 only. There will be a follow-up 12 weeks after the end of the trials. This follow-up will assess online questionnaires about physical and psychological well-being.

The objectives of this project are:

* To evaluate the effectiveness of HIFT, Qigong and MBSR interventions on the cognitive and psychological well-being of college students.
* To study the intervention-induced changes in the microbiome and brain structure and function (volume of gray and white matter, microstructural integrity, functional connectivity) and their potential mediator effect on cognitive and psychological well-being outcomes.
* To study the intervention-induced changes in the physical (physical activity and fitness status), mental (mindful thinking, sleep quality, and fatigue), and physiological stress (HRV) components and their potential mediator effect on cognitive and psychological well-being outcomes.
* To determine the potential moderator effects of demographic (sex, age and educational level) and individual factors (cognitive reserve, general intelligence) with intervention-induced changes in cognitive and psychological well-being outcomes.

In addition, the Study 2 also has these objectives:

* To generate the virtual environment of the designed interventions (HIFT-VR, Qigong-VR, and MBSR-VR).
* To evaluate the usability, acceptability, and outcomes of the newly developed VR interventions in relation to cognitive and emotional health to explore the feasibility of each VR intervention.
* To study the intervention-induced changes in the physical (physical activity and fitness status), mental (mindful thinking and sleep quality) and physiological stress (HRV) components and their potential mediator effect.
* To compare effects and adherences of traditional versus VR-based interventions.

ELIGIBILITY:
Inclusion Criteria:

* Individuals aged 18-25 years old
* Fluency in Catalan or Spanish (I.e., able to understand and speak)
* Accept to take part in the study and sign the informed consent according to the Declaration of Helsinki.

Exclusion Criteria:

* Severe Neurological or psychiatric history
* Alcohol or drug abuse history
* Injury that prevents exercise

Exclusion criteria only for MRI examination:

* Claustrophobia
* Medical device (e.g., pacemaker implants, stents)
* Other metal objects in the body

Exclusion criteria only for VR study:

* Dizziness
* Contraindications or troubles that could condition the use of VR

Ages: 18 Years to 25 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 219 (Estimated)
Dates: Start 2023-12-20 (Actual); Primary Completion 2026-05-18 (Estimated); Study Completion 2026-09-18 (Estimated)

PRIMARY OUTCOMES:
Changes in immediate verbal attention | Baseline (2 weeks before) & follow-up (2 weeks after completing interventions)
  Direct Digit Span, subtest from the Wechsler Adult Intelligence Scale - Third Edition (WAIS-III). Span. Direct score. Range 0-9. Higher scores indicate better performance.
Changes in processing speed | Baseline (2 weeks before) & follow-up (2 weeks after completing interventions)
  Symbol-Digit Coding subtest from the Wechsler Adult Intelligence Scale - Third Edition (WAIS-III). Direct score. Range 0-133. Higher scores indicate better performance.
Changes in visual attention | Baseline (2 weeks before) & follow-up (2 weeks after completing interventions)
  Trail Making Test Part A. Seconds to complete the numerical sequence. Direct score. More time indicates worse performance.
Changes in verbal memory | Baseline (2 weeks before) & follow-up (2 weeks after completing interventions)
  Rey Auditory Verbal Learning Test. Direct score. Range 0-75. Higher scores indicate better performance.
Changes in visual memory | Baseline (2 weeks before) & follow-up (2 weeks after completing interventions)
  Rey-Osterrieth Complex Figure. The memory drawing accuracy at 3-5 minutes. Direct score. Range 0-36. Higher scores indicate better performance.
Changes in Executive Function - Flexibility | Baseline (2 weeks before) & follow-up (2 weeks after completing interventions)
  Trail Making Test Part B. Seconds to complete the alphanumeric sequence. Direct score. More time indicates worse performance.
Changes in Executive Function - Inhibition | Baseline (2 weeks before) & follow-up (2 weeks after completing interventions)
  Stroop Color and Word Test. Interference of the Stroop Color and Word Test. Interference is calculated as follows: CW - ((W * C) / (W + C)). Higher scores indicate better performance. Negative values are possible, meaning a bad performance.
Changes in Executive Function - Verbal Fluency | Baseline (2 weeks before) & follow-up (2 weeks after completing interventions)
  Phonetic Fluency is measured using the Controlled Oral Word Association Test, spanish adaptation, and semantic fluency test using the category Animal. The total number of evoked words starting with the letters P, M, and R (60 seconds for each letter) and animals (60 seconds). Direct score. Higher scores indicate better performance.
Change in verbal digit working memory | Baseline (2 weeks before) & follow-up (2 weeks after completing interventions)
  Backward Digit Span subtest from the Wechsler Adult Intelligence Scale - Third Edition (WAIS-III). Span. Direct score. Range 0-8. Higher scores indicate better performance.
Changes in Verbal Comprehension | Baseline (2 weeks before)
  Vocabulary subtest from the Wechsler Adult Intelligence Scale - Third Edition (WAIS-III). Direct score. Range 0-66. Higher scores indicate better performance.
Changes in Psychological symptoms | Baseline (2 weeks before) & follow-up (2 weeks after completing interventions)
  90 Symptoms Inventory (90-SCL-R). Direct scores from 0 to 4. Higher scores indicate more symptomatology.
Changes in Self-esteem | Baseline (2 weeks before) & follow-up (2 weeks after completing interventions)
  Rosenberg Self-esteem scale (RSE). Direct scores from 10 to 40. Higher scores indicate higher self-esteem.
Changes in Depression, anxiety and stress | Baseline (2 weeks before) & follow-up (2 weeks after completing interventions)
  Depression, Anxiety and Stress Scale-21 (DASS-21). Direct score. Range 0-126. Higher scores indicate more global symptoms
Changes in Mindfulness | Baseline (2 weeks before) & follow-up (2 weeks after completing interventions)
  Five facet mindfulness questionnaire (FFMQ). Direct scores from 39 to 195. Higher scores indicate more Mindfulness levels.
Changes in Self-efficacy | Baseline (2 weeks before) & follow-up (2 weeks after completing interventions)
  General self-efficacy scale (GSE). Direct scores from 10 to 40. Higher scores indicate more self-eficacy.
Changes in Sleep quality | Baseline (2 weeks before) & follow-up (2 weeks after completing interventions)
  Pittsburgh Sleep Quality Index (PSQI). Direct score. Range 0-21. Lower scores indicate better sleep quality.
Changes in Diet | Baseline (2 weeks before) & follow-up (2 weeks after completing interventions)
  Mediterranean Diet Assessment Tool (PREDIMED). Direct score. Range 0-14. Higher scores indicate more adherence to a Mediterranean diet.

SECONDARY OUTCOMES:
Changes in Physical activity | Baseline (2 weeks before) & follow-up (2 weeks after completing interventions)
  International Physical Activity Questionnaire (IPAQ). Total physical activity measured in MET-min/week through the International Physical Activity Questionnaire - Short Form. Direct score. Higher scores indicate more physical activity.
Changes in Anthropometric Measurements - Height | Baseline (2 weeks before) & follow-up (2 weeks after completing interventions)
  Height in meters
Changes in Anthropometric Measurements - Weight | Baseline (2 weeks before) & follow-up (2 weeks after completing interventions)
  Weight in Kg
Changes in Anthropometric Measurements - Body Mass | Baseline (2 weeks before) & follow-up (2 weeks after completing interventions)
  Body mass index (BMI)
Changes in Anthropometric Measurements - Waist and hip circumference | Baseline (2 weeks before) & follow-up (2 weeks after completing interventions)
  Waist and hip circumference. Waist-to-hip ratio.
Changes in Physiological stress - Heart rate variability | Baseline (2 weeks before) & follow-up (2 weeks after completing interventions)
  RMSSD
Changes in Physiological stress - blood pressure | Baseline (2 weeks before) & follow-up (2 weeks after completing interventions)
  Blood pressure. Sistolic and diastolic blood pressure in millimeters of mercury.
Changes in aerobic capacity | Baseline (2 weeks before) & follow-up (2 weeks after completing interventions)
  Submaximal oxygen consumption test. Estimated VO2 score from submaximal step test.
Changes in lower body muscle power | Baseline (2 weeks before) & follow-up (2 weeks after completing interventions)
  Countermovement jump. Initial velocity and power output in countermovement jump in meters per second.
Changes in strength of the hand flexor muscles | Baseline (2 weeks before) & follow-up (2 weeks after completing interventions)
  Han-grip test. Right and left hand grip strength in kilogram-force.
Changes in balance | Baseline (2 weeks before) & follow-up (2 weeks after completing interventions)
  Y-balance test. Composite score of left leg Y Balance Test (% of leg length) (in cm). Formula = ((YBALANCE_L_ANTERIOR + YBALANCE_L_POSTEROMEDIAL + YBALANCE_L_POSTEROLATERAL) / (3 * LEG_LENGTH)) * 100
Changes in flexibility | Baseline (2 weeks before) & follow-up (2 weeks after completing interventions)
  Sit-and-reach test. Corrected sit and reach distance in centimeters.
Changes in White matter integrity | Baseline (2 weeks before) & follow-up (2 weeks after completing interventions)
  White matter integrity: tractography
Changes in Resting-state connectivity | Baseline (2 weeks before) & follow-up (2 weeks after completing interventions)
  Resting state brain activity using fMRI
Changes in brain volumetry | Baseline (2 weeks before) & follow-up (2 weeks after completing interventions)
  Grey and white matter volume measured by MRI
Microbiota data | Baseline (2 weeks before) & follow-up (2 weeks after completing interventions)
  Quantification of different bacterial species from the fresh stool samples
Changes in emotional status | Follow-up (2 weeks after completing interventions)
  Semi-structured interview with qualitative content and sentiment analysis
Usability Virtual Reality System: | Follow-up (2 weeks after completing interventions)
  System Usability Scale (SUS). Direct scores from 0 to 100. Higher scores indicate more usability

CONTACTS AND LOCATIONS:
Overall Officials: Maria Mataró, PhD, Principal Investigator — University of Barcelona
Locations (1):
- Maria Mataro, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Rostami S, Bermudo-Gallaguet A, Camins-Vila N, Ferrer-Uris B, Busquets A, Ribera M, Coll L, Gallego Vila J, Oliva Martinez R, Slater M, Garcia Diez G, Perales Castellanos N, Larrosa M, Bielsa-Pascual J, Toran-Montserrat P, Bruna Rabassa O, Guerra-Balic M, Erickson KI, Brown B, Serrat MM. The YoungFitT project: Study protocol for a randomized mixed-methods trial of physical exercise and mind-body interventions, with or without virtual reality, in university students. PLoS One. 2025 Aug 1;20(8):e0328538. doi: 10.1371/journal.pone.0328538. eCollection 2025. PMID 40748900